CLINICAL TRIAL: NCT03215030
Title: A Phase 1/2 Open-label Study to Investigate the Safety and Tolerability, Efficacy, Pharmacokinetics, and Immunogenicity of Modakafusp Alfa (TAK-573) as a Single Agent in Patients With Relapsed Refractory Multiple Myeloma
Brief Title: A Study of Modakafusp Alfa on Adult Participants With Relapsed/Refractory Multiple Myeloma
Acronym: iinnovate-1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated by the sponsor for strategic reasons
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-573-1501; TV48573-ONC-10128 (Other: Former Id); U1111-1195-8134 (Registry Identifier: WHO); 2021-006038-37 (EudraCT Number); jRCT2061220078 (Registry Identifier: jRCT)
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part 1 (Dose Escalation) Schedule A (Experimental): Participants received Modakafusp alfa 0.001 up to 0.75 milligram per kilogram (mg/kg), infusion, intravenously (IV), once every week (Q1W) on Days 1, 8, 15 and 22 of each 28-day treatment cycle up to 2 cycles, followed by once every 2 weeks (Q2W) on Days 1 and 15 of each 28-day treatment cycle up to 4 cycles, followed by once every 4 weeks (Q4W) on Day 1 of each 28-day treatment cycle until treatment discontinuation.
  Interventions: Drug: Modakafusp alfa
- Part 1 (Dose Escalation) Schedule B (Experimental): Participants received Modakafusp alfa 0.20 up to 0.30 mg/kg, infusion, IV, Q2W on Days 1 and 15 of each 28-day treatment cycle until treatment discontinuation.
  Interventions: Drug: Modakafusp alfa
- Part 1 (Dose Escalation) Schedule C (Experimental): Participants received Modakafusp alfa 0.40 up to 0.75 mg/kg, infusion, IV, once every 3 weeks (Q3W) on Day 1 of each 21-day treatment cycle until treatment discontinuation.
  Interventions: Drug: Modakafusp alfa
- Part 1 (Dose Escalation) Schedule D (Experimental): Participants received Modakafusp alfa 1.5 up to 6.0 mg/kg, infusion, IV, Q4W on Day 1 of each 28-day treatment cycle until treatment discontinuation.
  Interventions: Drug: Modakafusp alfa
- Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa (Experimental): Participants received modakafusp alfa 0.400 mg/kg infusion, IV, Q3W on Day 1 of each 21-day treatment cycle until treatment discontinuation.
  Interventions: Drug: Modakafusp alfa
- Part 2 (Dose Expansion):ScheduleC:Modakafusp Alfa+Dexamethasone (Experimental): Participants received modakafusp alfa 0.400 mg/kg infusion, IV, and dexamethasone 40 mg, orally, Q3W on Day 1 of each 21-day treatment cycle until treatment discontinuation.
  Interventions: Drug: Modakafusp alfa; Drug: Dexamethasone
- Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa (Experimental): Participants received modakafusp alfa 1.500 mg/kg infusion, IV, Q4W on Day 1 of each 28-day treatment cycle until treatment discontinuation.
  Interventions: Drug: Modakafusp alfa
- Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone (Experimental): Participants received modakafusp alfa 1.500 mg/kg infusion, IV, and dexamethasone 40 mg, orally, Q4W on Day 1 of each 28-day treatment cycle until treatment discontinuation.
  Interventions: Drug: Modakafusp alfa; Drug: Dexamethasone
- Part 3 (Dose Extension): Modakafusp Alfa 120 mg (Experimental): Participants received modakafusp alfa 120 mg, infusion, IV, Q4W, for each 28-day treatment cycle until disease progression or treatment discontinuation.
  Interventions: Drug: Modakafusp alfa
- Part 3 (Dose Extension): Modakafusp Alfa 240 mg (Experimental): Participants received modakafusp alfa 240 mg, infusion, IV, Q4W, for each 28-day treatment cycle until disease progression or treatment discontinuation.
  Interventions: Drug: Modakafusp alfa
- Japan Lead-in: Modakafusp Alfa 60 mg (Experimental): Participants received modakafusp alfa 60 mg, infusion, IV, Q4W, for each 28-day treatment cycle until disease progression or treatment discontinuation.
  Interventions: Drug: Modakafusp alfa
- Japan Lead-in: Modakafusp Alfa 120 mg (Experimental): Participants received modakafusp alfa 120 mg, infusion, IV, Q4W, for each 28-day treatment cycle until disease progression or treatment discontinuation.
  Interventions: Drug: Modakafusp alfa

INTERVENTIONS:
Drug: Modakafusp alfa — Modakafusp alfa intravenous infusion.
  Other Names: TAK-573; TEV-48573
Drug: Dexamethasone — Dexamethasone.
  Arms: Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone; Part 2 (Dose Expansion):ScheduleC:Modakafusp Alfa+Dexamethasone

SUMMARY:
The main aims of this 3-part study are as follows:

Part 1: To determine any side effects from modakafusp alfa single treatment and how often they occur. The dose of modakafusp alfa will be increased a little at a time until the highest dose that does not cause harmful side effects is found.

Part 2: To assess clinical activity of one or more dosing schedules of modakafusp alfa alone in participants with relapsed/refractory multiple myeloma. Dexamethasone standard dose will be administered with one or more selected dose of modakafusp alfa in selected group of participants.

Part 3: To find the optimal dose with the more favorable risk-benefit profile of modakafusp alfa.

Participants will receive modakafusp alfa at one of two doses which will be given through a vein.

DETAILED DESCRIPTION:
The drug being tested in this study, and which will be given through a vein, is called modakafusp alfa (TAK-573 ) as single agent or in combination with dexamethasone. The study will determine the safety, tolerability, and efficacy of modakafusp alfa as single agent and in combination with dexamethasone in participants with relapsed/refractory multiple myeloma (RRMM). The study consists of 3 Parts:

Part 1: Dose Escalation, Part 2: Dose Expansion, Part 3: Dose Extension

The study will enroll approximately 65 participants in Part 1, 35 in Part 2, and 236 in Part 3. Participants will be assigned to one of the following treatment groups in Parts 1 and 2 of the study. Participants will be randomly assigned in Part 3 of the study as given below:

* Part 1 (Dose Escalation) Schedule A: Modakafusp alfa 0.001 Up to 14 mg/kg
* Part 1 (Dose Escalation) Schedule B: Modakafusp alfa TBD
* Part 1 (Dose Escalation) Schedule C: Modakafusp alfa TBD
* Part 1 (Dose Escalation) Schedule D: Modakafusp alfa TBD
* Part 2 (Dose Expansion): Modakafusp alfa TBD + Dexamethasone 40 mg
* Part 3 (Dose Extension): Modakafusp alfa 120 mg
* Part 3 (Dose Extension): Modakafusp alfa 240 mg

The Part 1 (Dose Escalation) portion of the study will follow a 3+3 dose escalation design to evaluate once-weekly up to 4 different schedules of administration of modakafusp alfa starting at 0.001 mg/kg for dose limiting toxicity (DLT) evaluation and to determine the maximum tolerated dose (MTD) or an optimal biological dose (OBD) for assessments in Part 2.

The Part 2 (Dose Expansion) will further assess the safety profile of modakafusp alfa and its efficacy at MTD or OBD.

For Part 3 (Dose Extension) participants will be randomized 1:1 to receive single-agent modakafusp alfa 120 mg or 240 mg Q4W.

Parts 1 and 2 will be conducted at multiple centers in the United States. Part 3 will be conducted worldwide. The maximum treatment duration in this study is up to 12 months (Parts 1 and 2) or until disease progression (Part 3) and overall time to participate in the study is approximately up to 90 months. Participants with clinical benefit may continue treatment after sponsor approval.

ELIGIBILITY:
Inclusion Criteria:

For Parts 1 and 2:

1. Has MM defined by the IMWG criteria with evidence of disease progression and:

* In need of additional myeloma therapy as determined by the investigator.
* Has previously received at least 3 lines of myeloma therapy (for example, containing an Immunomodulatory imide drug [IMiD], a proteasome inhibitor [PI], an alkylating agent, and/or an anti-CD38 as single agents or in combination).
* Is either refractory to or intolerant of at least 1 PI and a least 1 IMiD.

For Part 3:

1. Has MM defined by the IMWG criteria with evidence of disease progression and:

   * In need of additional myeloma therapy as determined by the investigator.
   * Has previously received at least 3 lines of myeloma therapy.
   * Is refractory to at least 1 IMiD (ie, lenalidomide or pomalidomide [thalidomide excluded]), at least 1 PI (ie, bortezomib, ixazomib, or carfilzomib), and refractory to at least 1 anti-CD38 antibody (ie, daratumumab or isatuximab) and has demonstrated disease progression with the last therapy. Participants who are primary refractory, meaning they never achieved at least a MR with any previous treatment line, are not eligible.
2. For participants in Part 2 and 3 only: Measurable disease is defined as :

   1. Serum M-protein ≥500 mg/dL (≥5 g/L)
   2. Urine M-protein ≥200 mg/24 hours.
   3. Serum free light chain (FLC) assay, with involved FLC level ≥10 mg/dL (≥100 mg/L) provided serum FLC ratio is abnormal.
3. During Part 1 only, participants not meeting the above criteria for measurable disease should, at least, have measurable bone marrow plasmacytosis (greater than or equal to [≥ ] 10 percent [%]) and/or plasmacytoma (≥1 centimeter [cm] in diameter) detected by physical examination or imaging.
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.

Exclusion Criteria:

For Parts 1 and 2:

1. Has polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes (POEMS) syndrome, monoclonal gammopathy of unknown significance, smoldering myeloma, solitary plasmacytoma, amyloidosis, Waldenstrom macroglobulinemia or immunoglobulin M (IgM) myeloma, or lymphoplasmacytic lymphoma (LPL).
2. Who have received autologous stem cell transplant (SCT) 60 days before first infusion of modakafusp alfa or participants who have received allogeneic SCT 6 months before first infusion. Graft-versus-host disease that is active or requires ongoing systemic immunosuppression.
3. Has not recovered from adverse reactions to prior myeloma treatment or procedures (chemotherapy, immunotherapy, radiation therapy) to NCI CTCAE less than or equal to (≤) Grade 1 or baseline, except for sensory or motor neuropathy which should have recovered to ≤ Grade 2 or baseline.
4. Has clinical signs of central nervous system involvement of MM.

For Part 3:

* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]. Participants with resolved infection (that is, participants who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of HBV DNA levels. Those who are PCR positive will be excluded.
* In addition to the above criteria, participants must not have plasma cell leukemia or have had primary refractory MM, current central nervous system involvement of MM, myelodysplastic syndrome, myeloproliferative syndrome, or have had a second malignancy within the previous 3 years, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, cervical carcinoma in situ, resected colorectal adenomatous polyps, breast cancer in situ, or other malignancy for which the participant is not on active anticancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (94):
- United States (27):
  - Highlands Oncology Group, Springdale, Arkansas
  - Los Angeles Cancer Network - Glendale Adventist Medical Center, Glendale, California
  - University of California Irvine, Orange, California
  - Office of James R. Berenson MD, West Hollywood, California
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwestern Medicine - Northwestern Medical Group, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Investigative Clinical Research of Indiana, LLC, Noblesville, Indiana
  - June E. Nylen Cancer Center, Sioux City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Univeristy of Nebraska Medical Center, Omaha, Nebraska
  - USOR - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - John Theurer Cancer Center, Hackensack, New Jersey
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Center, Charlotte, North Carolina
  - Levine Cancer Institute - Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baptist Cancer Center - Memphis - Walnut Grove, Memphis, Tennessee
  - Lumi Research, Houston, Texas
- Canada (4):
  - British Columbia Cancer Agency Vancouver Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Centre de Recherche du CHUM, Montreal, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
- China (11):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University - Suzhou First People's Hospital, Suzhou, Jiangsu
  - Shanghai Fourth People's Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
- France (10):
  - Institut de cancerologie Strasbourg Europe, Strasbourg, Alsace
  - Hopital Saint-Vincent de Paul - Lille, Lille, Hauts-de-France
  - Centre Hospitalier Regional Universitaire de Lille, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire de Toulouse Hopital Purpan, Toulouse, Midi-pyrenees
  - Centre Hospitalier Universitaire Nantes - Hotel Dieu, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Poitiers, Poitiers, Poitou-charentes
  - Centre Hospitalier d'Argenteuil - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier Universitaire Henri Mondor, Créteil, Île-de-France Region
  - Hopital Saint-Antoine, Paris, Île-de-France Region
  - Hopital Necker-Enfants Malades, Paris, Île-de-France Region
- Germany (2):
  - Universitatsklinik Tubingen, Tübingen, Baden-Wurttemberg
  - Universitatsklinikum Leipzig, Leipzig, Saxony
- Greece (3):
  - Evaggelismos General Hospital, Athens, Attica
  - Alexandra General Hospital of Athens, Athens, Attica
  - University Regional General Hospital of Patras, Patra, Peloponnese
- Israel (3):
  - The Chaim Sheba Medical Center, Ramat Gan, Tel Aviv
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (5):
  - AON SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico Sant'Orsola-Malpighi, Bologna
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele, Catania
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Japan (5):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Ogaki Municipal Hospital, Gifu, Gifu
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - Japanese Red Cross Medical Center, Tokyo
- Oslo Universitetssykehus-Ulleval Hospital, Oslo, Norway
- Puerto Rico (2):
  - Ad-Vance Medical Research, Ponce, PR
  - Hospital Espanol Auxilio Mutuo, San Juan
- South Korea (3):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea - Seoul St. Mary's Hospital, Seoul
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
- Taiwan (2):
  - Tri-Service General Hospital, Taipei, Taipei CITY
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (2):
  - Ankara Universitesi, Yenimahalle, Ankara
  - Ondokuz Mayis Universitesi Tp Fakultesi, Samsun
- United Kingdom (7):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, England
  - Royal Cornwall Hospital NHS Trust, Cornwell, England
  - University College London Hospitals NHS Foundation Trust, London, England
  - Genesis Care - Milton Keynes, Milton Keynes, England
  - Oxford University Hospitals NHS Foundation Trust, Oxford, England
  - The Royal Marsden NHS Foundation Trust, Sutton, England
  - Genesis Care Windsor - Genesis Care UK Ltd., Windsor, England

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please visit USMedInfo@tevapharm.com to make your request.

REFERENCES:
- [Derived] Holstein SA, Atrash S, Mian H, Dimopoulos MA, Schjesvold F, Popat R, Shah N, Gatt ME, Gocke CB, Frenzel L, Touzeau C, Beksac M, Manier S, Magen H, Travis P, Nadeem O, Suryanarayan K, Li C, Li S, Nelson A, Cherepanov D, Parot X, Vogl DT. A phase 2 randomized study of modakafusp alfa as a single agent for patients with relapsed/refractory multiple myeloma. Blood. 2025 Aug 28;146(9):1051-1064. doi: 10.1182/blood.2024027873. PMID 40279508
- [Derived] Vogl DT, Atrash S, Holstein SA, Nadeem O, Benson D, Chaudry M, Biran N, Suryanarayan K, Li C, Liu Y, Collins S, Parot X, Kaufman JL. Targeted interferon therapy with modakafusp alfa for relapsed or refractory multiple myeloma. Blood. 2025 Feb 27;145(9):944-955. doi: 10.1182/blood.2024026124. PMID 39630057

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 4 October 2017 to 7 November 2024.
Pre-assignment Details: Participants with diagnosis of RRMM were enrolled in this study consisting of Part 1 (Dose Escalation), Part 2 (Dose Expansion), Part 3 (Dose Extension), & Japan Safety Lead-in to receive modakafusp alfa with/without dexamethasone. 4 participants enrolled in study but discontinued without receiving TAK-573 dosing and are thus not presented below.
Groups:
- Part2(Dose Expansion):ScheduleC:Modakafusp Alfa+Dexamethasone: Participants received modakafusp alfa 0.400 mg/kg infusion, IV, and dexamethasone 40 mg, orally, Q3W on Day 1 of each 21-day treatment cycle until treatment discontinuation.
Period: Part 1: Dose Escalation
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part2(Dose Expansion):ScheduleC:Modakafusp Alfa+Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg | Japan Lead-in: Modakafusp Alfa 60 mg | Japan Lead-in: Modakafusp Alfa 120 mg
Started | 20 | 8 | 7 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 1 | 1 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 18 | 7 | 6 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 15 | 6 | 6 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Dose Expansion
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part2(Dose Expansion):ScheduleC:Modakafusp Alfa+Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg | Japan Lead-in: Modakafusp Alfa 60 mg | Japan Lead-in: Modakafusp Alfa 120 mg
Started | 0 | 0 | 0 | 0 | 8 | 3 | 25 | 25 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 4 | 1 | 11 | 16 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 4 | 2 | 14 | 9 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 3 | 1 | 5 | 4 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0
Period: Part 3: Dose Extension
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part2(Dose Expansion):ScheduleC:Modakafusp Alfa+Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg | Japan Lead-in: Modakafusp Alfa 60 mg | Japan Lead-in: Modakafusp Alfa 120 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 71 | 75 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 66 | 68 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 38 | 39 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 7 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 20 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Period: Japan Safety Lead-In
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part2(Dose Expansion):ScheduleC:Modakafusp Alfa+Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg | Japan Lead-in: Modakafusp Alfa 60 mg | Japan Lead-in: Modakafusp Alfa 120 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Parts 1 and 2: The Safety Analysis Set (SAS) included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573.
  Part 3 and Japan Lead-in: The Full Analysis Set (FAS) included all enrolled participants who received at least 1 dose of study drug even if dose was incomplete.
Groups:
- Part 1 (Dose Escalation) Schedule A: Participants received modakafusp alfa 0.001 up to 0.75 mg/kg, infusion, IV, Q1W on Days 1, 8, 15 and 22 of each 28-day treatment cycle up to 2 cycles, followed by Q2W on Days 1 and 15 of each 28-day treatment cycle up to 4 cycles, followed by Q4W on Day 1 of each 28-day treatment cycle until treatment discontinuation.
- Part 1 (Dose Escalation) Schedule C: Participants received modakafusp alfa 0.40 up to 0.75 mg/kg, infusion, IV, Q3W on Day 1 of each 21-day treatment cycle until treatment discontinuation.
- Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone: Participants received modakafusp alfa 0.400 mg/kg infusion, IV, and dexamethasone 40 mg, orally, Q3W on Day 1 of each 21-day treatment cycle until treatment discontinuation.
- Total: Total of all reporting groups
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg | Japan Lead-in: Modakafusp Alfa 60 mg | Japan Lead-in: Modakafusp Alfa 120 mg | Total
Number analyzed (Participants) | 20 | 8 | 7 | 21 | 8 | 3 | 25 | 25 | 71 | 75 | 3 | 2 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.56) | 61.1 (7.00) | 60.4 (10.47) | 64.7 (10.34) | 61.9 (8.63) | 65.7 (12.58) | 64.1 (12.17) | 70.2 (7.77) | 66.2 (9.76) | 66.5 (9.61) | 66.66 (9.71) | 66.00 (11.31) | 65.46 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 2 | 10 | 1 | 2 | 12 | 10 | 34 | 39 | 2 | 0 | 125
  Male | 10 | 5 | 5 | 11 | 7 | 1 | 13 | 15 | 37 | 36 | 1 | 2 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 0 | 0 | 10
  Not Hispanic or Latino | 19 | 8 | 6 | 21 | 8 | 3 | 24 | 23 | 51 | 57 | 3 | 2 | 225
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 16 | 15 | 0 | 0 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 5 | 9 | 3 | 2 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 1 | 5 | 1 | 0 | 2 | 8 | 10 | 4 | 0 | 0 | 34
  White | 20 | 4 | 6 | 14 | 6 | 3 | 20 | 17 | 38 | 51 | 0 | 0 | 179
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 18 | 11 | 0 | 0 | 32

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants Reporting One or More Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participants administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. A TEAE is defined as any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last administration of study drug.
Time Frame: Up to 54.3 months in Part 1
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D
Number analyzed (Participants) | 20 | 8 | 7 | 21
percentage of participants | 100 | 100 | 100 | 100

2. Primary Outcome: Part 1: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs were evaluated as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0. Nonhematologic TEAEs of NCI CTCAE Grade ≥3 clearly unrelated to the underlying disease and occurring during the first cycle were considered DLTs.
Time Frame: Up to Cycle 1 (cycle length was 28 days for Schedule A, B and D; 21 days for Schedule C)
Population: The DLT-evaluable Analysis Set included participants who received all Cycle 1 doses of modakafusp alfa or experienced a DLT in Cycle 1 in the Part 1 Dose Escalation portion of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D
Number analyzed (Participants) | 13 | 6 | 7 | 21
Participants | 4 | 3 | 0 | 3

3. Primary Outcome: Part 1: Percentage of Participants Reporting One or More Grade 3 or Higher TEAEs
Description: An AE is defined as any untoward medical occurrence in a participants administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. TEAEs grades were evaluated as per NCI CTCAE, Version 5.0. Grade 1 scaled as mild; Grade 2 scaled as moderate; Grade 3 scaled as severe or medically significant but not immediately life-threatening; Grade 4 scaled as life-threatening consequences; and Grade 5 scaled as death related to AE. Percentages were rounded off to the nearest decimal.
Time Frame: Up to 54.3 months in Part 1
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D
Number analyzed (Participants) | 20 | 8 | 7 | 21
percentage of participants | 95 | 100 | 85.7 | 95.2

4. Primary Outcome: Part 1: Percentage of Participants Reporting One or More Serious Treatment-emergent Adverse Events (Serious TEAEs)
Description: AE: any untoward medical occurrence in participants administered a pharmaceutical product; untoward medical occurrence does not necessarily have causal relationship with this treatment. AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of medicinal (investigational) product whether or not it is related to medicinal product. TEAE: any AE either reported for first time or worsening of pre-existing event after first dose of study drug & within 30 days of last administration of study drug. Serious TEAEs: any untoward medical occurrence that: 1)results in death, 2) is life-threatening, 3) requires inpatient hospitalization or prolongation of existing hospitalization, 4) results in persistent or significant disability/incapacity, 5) leads to a congenital anomaly/birth defect in the offspring of the participant or 6) is medically important event. Percentages were rounded off to nearest decimal.
Time Frame: Up to approximately 54.3 months in Part 1
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D
Number analyzed (Participants) | 20 | 8 | 7 | 21
percentage of participants | 40 | 75 | 28.6 | 61.9

5. Primary Outcome: Part 1: Percentage of Participants Who Discontinued the Treatment Because of TEAE
Description: An AE is defined as any untoward medical occurrence in a participants administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. A TEAE is defined as any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last administration of study drug. Percentages were rounded off to the nearest decimal.
Time Frame: Up to 54.3 months in Part 1
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D
Number analyzed (Participants) | 20 | 8 | 7 | 21
percentage of participants | 15 | 25 | 0 | 14.3

6. Primary Outcome: Part 1: Percentage of Participants With TEAEs Resulting in Dose Modifications: Dose Delay
Description: Percentages were rounded off to the nearest decimal.
Time Frame: Up to 54.3 months in Part 1
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D
Number analyzed (Participants) | 20 | 8 | 7 | 21
percentage of participants | 30 | 12.5 | 57.1 | 9.5

7. Primary Outcome: Part 1: Percentage of Participants With TEAEs Resulting in Dose Modifications: Dose Interruptions
Description: Percentages were rounded off to the nearest decimal.
Time Frame: Up to 54.3 months in Part 1
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D
Number analyzed (Participants) | 20 | 8 | 7 | 21
percentage of participants | 15 | 0 | 0 | 0

8. Primary Outcome: Part 1: Percentage of Participants With TEAEs Resulting in Dose Modifications: Dose Reductions
Description: Percentages were rounded off to the nearest decimal.
Time Frame: Up to 54.3 months in Part 1
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D
Number analyzed (Participants) | 20 | 8 | 7 | 21
percentage of participants | 10 | 12.5 | 0 | 9.5

9. Primary Outcome: Part 1: Percentage of Participants With Clinically Significant Laboratory Values
Description: Laboratory values included hematology, chemistry, and urinalysis and were assessed per investigator's interpretation.
Time Frame: Up to 54.3 months in Part 1
Population: SAS:all participants who took ≥1 dose,even if incomplete,of TAK-573.However,clinically significant laboratory values data were not collected & will never be available to present due to an issue with report form used for data collection(identified after trial completion).Assessments of clinical significance were not included in the report form,making data collection impossible.This issue did not impact participant safety or reliability of study data,particularly primary endpoint.
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Primary Outcome: Part 1: Percentage of Participants With Clinically Significant Vital Signs Measurements
Description: Vital signs included temperature, pulse, respiratory rate, oxygen saturation, and blood pressure.
Time Frame: Up to 54.3 months in Part 1
Population: SAS:all participants who took ≥1 dose,even if incomplete,of TAK-573.However,clinically significant vital signs measurements data were not collected & will never be available to present due to an issue with report form used for data collection(identified after trial completion).Assessments of clinical significance were not included in the report form,making data collection impossible.This issue did not impact participant safety or reliability of study data,particularly primary endpoint.
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Primary Outcome: Part 2: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved a partial response (PR) rate or better (stringent complete response [sCR] + complete response [CR] + very good partial response [VGPR] + PR) during the study as defined by international myeloma working group (IMWG) uniform response criteria. PR: ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. CR: negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow. sCR: CR+normal free light chain (FLC) ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry. VGPR:serum and urine M-protein detectable by immunofixation but not on electrophoresis, or ≥90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours.
Time Frame: Up to 34.7 months in Part 2
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573 and with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone
Number analyzed (Participants) | 8 | 3 | 25 | 25
percentage of participants | 0 [0.00 to 36.94] | 0 [0.00 to 70.76] | 48 [27.80 to 68.69] | 32 [14.95 to 53.50]

12. Primary Outcome: Part 3: Overall Response Rate (ORR) Assessed by Independent Review Committee (IRC)
Description: ORR was defined as the percentage of participants who achieved a PR rate or better (sCR + CR + VGPR + PR) during the study as defined by IMWG uniform response criteria. PR :≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. CR:negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow. Scr: CR+normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry. VGPR:serum and urine M-protein detectable by immunofixation but not on electrophoresis, or ≥90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours.
Time Frame: Up to 20.5 months in Part 3
Population: The FAS included all participants who received at least 1 dose, even an incomplete dose, of modakafusp alfa, in the Part 3 extension cohorts. Due to early termination, IRC was disbanded prior to completing its evaluation and could not be utilized for the assessment, therefore the data for this outcome measure is not available.
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Dose-limiting Toxicities (DLTs)- Like Events
Description: Percentage of participants with TEAEs meeting DLT definition were reported. Toxicity was evaluated as per the NCI CTCAE, Version 5.0. The hematologic TEAEs of Grade ≥3 clearly unrelated to the underlying disease and occur during the first cycle that are considered DLTs: Grade ≥3 hemolysis; Grade 4 neutropenia for >7 consecutive days; Grade 4 thrombocytopenia for >14 consecutive days; Grade 3 thrombocytopenia with clinically significant bleeding; Any other Grade ≥4 hematologic toxicity except for Grade 4 lymphopenia. An incomplete recovery from treatment-related toxicity causing >2-week delay in the next scheduled infusion before the initiation of Cycle 2 were considered a DLT. Percentages were rounded off to the nearest decimal.
Time Frame: Up to 54.3 months in Part 1; Up to 34.7 months in Part 2
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone
Number analyzed (Participants) | 20 | 8 | 7 | 21 | 8 | 3 | 25 | 8
percentage of participants | 10 | 0 | 0 | 9.5 | 12.5 | 66.7 | 24 | 25

14. Secondary Outcome: Part 1: Cmax: Maximum Observed Serum Concentration for Modakafusp Alfa
Description: As per planned analysis, data for this outcome measure was collected and reported dose-wise for each treatment schedule.
Time Frame: Part 1:Schedule A:Day 1&15 in Cycles 1&2; Schedule B: Day1&15 in Cycles 1&2; Schedule C:Day1 in Cycles 1&2; Schedule D: Day 1 in Cycles 1&2: Pre-infusion&at multiple times post-infusion (cycle length was 28 days for Schedule A, B&D;21 days for Schedule C)
Population: The Pharmacokinetic (PK) Analysis Set included participants from the SAS who had sufficient data to calculate at least 1 PK parameter for modakafusp alfa. Overall number of participants analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis during the specified time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.01 mg/kg: Participants received modakafusp alfa 0.01 mg/kg, infusion, IV, Q1W on Days 1, 8, 15 and 22 of each 28-day treatment cycle up to 2 cycles, followed by once on Days 1 and 15 of each 28-day treatment cycle up to 4 cycles, followed by once on Day 1 of each 28-day treatment cycle until treatment discontinuation.
- Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.1 mg/kg: Participants received modakafusp alfa 0.1 mg/kg, infusion, IV, Q1W on Days 1, 8, 15 and 22 of each 28-day treatment cycle up to 2 cycles, followed by once on Days 1 and 15 of each 28-day treatment cycle up to 4 cycles, followed by once on Day 1 of each 28-day treatment cycle until treatment discontinuation.
- Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.4 mg/kg: Participants received modakafusp alfa 0.4 mg/kg, infusion, IV, Q1W on Days 1, 8, 15 and 22 of each 28-day treatment cycle up to 2 cycles, followed by once on Days 1 and 15 of each 28-day treatment cycle up to 4 cycles, followed by once on Day 1 of each 28-day treatment cycle until treatment discontinuation.
- Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.75 mg/kg: Participants received modakafusp alfa 0.75 mg/kg, infusion, IV, Q1W on Days 1, 8, 15 and 22 of each 28-day treatment cycle up to 2 cycles, followed by once on Days 1 and 15 of each 28-day treatment cycle up to 4 cycles, followed by once on Day 1 of each 28-day treatment cycle until treatment discontinuation.
- Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.2 mg/kg: Participants received Modakafusp alfa 0.2 mg/kg, infusion, IV, Q2W on Days 1 and 15 of each 28-day treatment cycle until treatment discontinuation.
- Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.3 mg/kg: Participants received modakafusp alfa 0.3 mg/kg, infusion, IV, Q2W on Days 1 and 15 of each 28-day treatment cycle until treatment discontinuation.
- Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.4 mg/kg: Participants received modakafusp alfa 0.4 mg/kg, infusion, IV, Q3W on Day 1 of each 21-day treatment cycle until treatment discontinuation.
- Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.75 mg/kg: Participants received modakafusp alfa 0.75 mg/kg, infusion, IV, Q3W on Day 1 of each 21-day treatment cycle until treatment discontinuation.
- Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 0.75 mg/kg: Participants received modakafusp alfa 0.75 mg/kg infusion, IV, Q4W on Day 1 of each 28-day treatment cycle until treatment discontinuation.
- Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 1.5 mg/kg: Participants received modakafusp alfa 1.5 mg/kg infusion, IV, Q4W on Day 1 of each 28-day treatment cycle until treatment discontinuation.
Arm/Group | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.01 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.1 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.2 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.3 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 1.5 mg/kg
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 4 | 4 | 4 | 2 | 6 | 3
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1 | 14.7 (47.6) | 154 (95.5) | 2980 (29.0) | 11800 (33.5) | 1260 (106.1) | 2230 (53.8) | 2460 (38.6) | 15000 (20.0) | 11600 (30.9) | 15900 (27.1)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 4 | 3 | 2 | 3 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 | 16.9 (75.4) | 289 (71.8) | 2750 (18.1) | 11900 (40.8) | 1030 (183.5) | 2600 (37.9) |  |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 1 | 3 | 2 | 5 | 2
  Cycle 2 Day 1 | 47.5 (175.1) | 158 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 3030 (10.1) |  |  | 1970 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 2490 (41.5) | 15100 (2.3) | 9690 (21.3) | 16800 (31.3)
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Cycle 2 Day 15 |  |  |  |  | 1730 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 1270 (NA) — Geometric coefficient of variation was not estimable for a single participant. |  |  |  |

15. Secondary Outcome: Part 1: Tmax: Time to Reach the Cmax for Modakafusp Alfa
Description: As per planned analysis, data for this outcome measure was collected and reported dose-wise for each treatment schedule.
Time Frame: as for outcome 14
Population: The PK Analysis Set included participants from the SAS who had sufficient data to calculate at least 1 PK parameter for modakafusp alfa. Overall number of participants analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis during the specified time-point.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.01 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.1 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.2 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.3 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 1.5 mg/kg
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 4 | 4 | 4 | 2 | 6 | 3
hours
  Cycle 1 Day 1 | 4.03 [3.97 to 4.15] | 3.99 [1.95 to 4.25] | 4.40 [3.92 to 6.10] | 4.27 [4.00 to 6.28] | 4.75 [3.97 to 5.60] | 4.03 [4.00 to 4.10] | 4.78 [3.87 to 6.05] | 3.07 [2.07 to 4.07] | 4.94 [4.00 to 6.02] | 4.03 [3.77 to 7.65]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 4 | 3 | 2 | 3 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 | 3.93 [2.02 to 4.05] | 4.02 [3.93 to 4.20] | 4.25 [4.08 to 4.35] | 5.87 [5.78 to 5.95] | 4.28 [4.15 to 6.17] | 4.00 [4.00 to 4.10] |  |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 1 | 3 | 2 | 5 | 2
  Cycle 2 Day 1 | 2.97 [1.97 to 3.98] | 4.23 [4.23 to 4.23] | 3.98 [3.90 to 4.05] |  |  | 4.45 [4.45 to 4.45] | 4.00 [3.90 to 5.92] | 3.21 [2.23 to 4.18] | 4.13 [3.90 to 5.95] | 5.52 [3.98 to 7.05]
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Cycle 2 Day 15 |  |  |  |  | 5.65 [5.65 to 5.65] | 4.00 [4.00 to 4.00] |  |  |  |

16. Secondary Outcome: Part 1: AUC∞: Area Under the Serum Concentration-time Curve From Time 0 to Infinity for Modakafusp Alfa
Description: As per planned analysis, data for this outcome measure was collected and reported dose-wise for each treatment schedule. Given the low exposure at the 0.1 mg/kg dose, there was insufficient data to characterize the terminal phase PK required for calculating this parameter. Consequently, this parameter has been marked as "Not Calculated" - and therefore not reported - for the Part 1, Schedule A, 0.1 mg/kg dose group, in accordance with non-compartmental PK analysis standards.
Time Frame: Part1:Schedule A:Day 1 in Cycles1&2&Day15 in Cycle1;Schedule B: Day1&15 in Cycle 1;Schedule C:Day1 in Cycles1&2; Schedule D:Day 1 in Cycles1&2: Pre-infusion&at multiple times post-infusion (cycle length= 28 days for Schedule A, B&D;21 days for Schedule C)
Population: PK Analysis Set; Overall number analyzed: participants with data available for analysis.Number analyzed: participants with data available during specified time-point.Given low exposure at 0.01mg/kg dose,there was insufficient data to characterize terminal phase PK required for calculating this parameter.Consequently,this parameter has been marked as "Not Calculated" and therefore not reported for Part 1,Schedule A,0.01mg/kg dose group,in accordance with non-compartmental PK analysis standards.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.01 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.1 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.2 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.3 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 1.5 mg/kg
Number analyzed (Participants) | 0 | 2 | 3 | 3 | 1 | 2 | 1 | 2 | 4 | 3
hour*nanogram per milliliter (h*ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 3 | 0 | 2 | 1 | 2 | 4 | 3
  Cycle 1 Day 1 |  |  | 14900 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 209000 (83.4) |  | 20500 (33.2) | 14100 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 288000 (44.5) | 199000 (104.4) | 240000 (109.7)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 2 | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 |  | 2410 (21.3) | 24000 (38.0) | 286000 (66.5) | 24300 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 20100 (21.7) |  |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 4 | 1
  Cycle 2 Day 1 |  |  | 28000 (49.3) |  |  |  | 73600 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 333000 (54.0) | 243000 (54.5) | 215000 (NA) — Geometric coefficient of variation was not estimable for a single participant.

17. Secondary Outcome: Part 1: AUClast: Area Under the Serum Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Modakafusp Alfa
Description: As per planned analysis, data for this outcome measure was collected and reported dose-wise for each treatment schedule.
Time Frame: as for outcome 16
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.01 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.1 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.2 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.3 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 1.5 mg/kg
Number analyzed (Participants) | 2 | 6 | 3 | 3 | 4 | 4 | 4 | 2 | 6 | 3
h*ng/mL
  Cycle 1 Day 1 | 29.5 (19.0) | 550 (111.6) | 30100 (67.9) | 208000 (83.2) | 7090 (263.7) | 10600 (98.0) | 17900 (106.8) | 287000 (44.5) | 197000 (83.9) | 229000 (107.7)
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 4 | 3 | 2 | 3 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 | 76.3 (34.8) | 1270 (88.4) | 23900 (38.2) | 285000 (66.1) | 8710 (514.0) | 19200 (17.0) |  |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 1 | 3 | 2 | 5 | 2
  Cycle 2 Day 1 | 128 (113.1) | 584 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 27700 (48.5) |  |  | 6020 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 15600 (225.4) | 332000 (54.0) | 190000 (77.5) | 582000 (250.5)
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Cycle 2 Day 15 |  |  |  |  | 22200 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 5090 (NA) — Geometric coefficient of variation was not estimable for a single participant. |  |  |  |

18. Secondary Outcome: Part 1: λz: Terminal Disposition Rate Constant for Modakafusp Alfa
Description: as for outcome 16
Time Frame: as for outcome 16
Population: PK Analysis Set; Overall number analyzed: participants with data available for analysis.Number analyzed: participants with data available during specified time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour (1/hour)
Arm/Group | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.01 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.1 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.2 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.3 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 1.5 mg/kg
Number analyzed (Participants) | 0 | 2 | 3 | 3 | 1 | 2 | 1 | 2 | 4 | 3
per hour (1/hour)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 3 | 0 | 2 | 1 | 2 | 4 | 3
  Cycle 1 Day 1 |  |  | 0.309 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 0.0933 (26.2) |  | 0.294 (3.1) | 0.265 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 0.0924 (0.5) | 0.107 (88.7) | 0.113 (117.8)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 2 | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 |  | 0.162 (4.3) | 0.207 (34.6) | 10.0852 (20.6) | 0.115 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 0.179 (59.7) |  |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 4 | 1
  Cycle 2 Day 1 |  |  | 0.197 (12.7) |  |  |  | 0.0907 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 0.0528 (10.1) | 0.0828 (14.6) | 0.0961 (NA) — Geometric coefficient of variation was not estimable for a single participant.

19. Secondary Outcome: Part 1: T1/2z: Terminal Elimination Phase Half-life for Modakafusp Alfa
Description: As per planned analysis, data for this outcome measure was collected and reported dose-wise for each treatment schedule.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.01 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.1 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.2 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.3 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 1.5 mg/kg
Number analyzed (Participants) | 0 | 2 | 3 | 3 | 1 | 2 | 1 | 2 | 4 | 3
hours
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 3 | 0 | 2 | 1 | 2 | 4 | 3
  Cycle 1 Day 1 |  |  | 2.24 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 7.43 (26.2) |  | 2.36 (3.1) | 2.61 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 7.50 (0.4) | 6.51 (88.6) | 6.16 (117.7)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 2 | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 |  | 4.28 (4.3) | 3.36 (34.6) | 8.14 (20.6) | 6.01 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 3.87 (59.7) |  |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 4 | 1
  Cycle 2 Day 1 |  |  | 3.52 (12.8) |  |  |  | 7.64 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 13.1 (10.1) | 8.37 (14.6) | 7.22 (NA) — Geometric coefficient of variation was not estimable for a single participant.

20. Secondary Outcome: Part 1: CL: Clearance for Modakafusp Alfa
Description: Clearance is defined as a quantitative measure of the rate at which a drug substance is removed from the body. CL = dose/AUC. As per planned analysis, data for this outcome measure was collected and reported dose-wise for each treatment schedule.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour per kilogram (L/h/kg)
Arm/Group | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.01 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.1 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.2 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.3 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 1.5 mg/kg
Number analyzed (Participants) | 0 | 2 | 3 | 3 | 1 | 2 | 1 | 2 | 4 | 3
liters per hour per kilogram (L/h/kg)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 3 | 0 | 2 | 1 | 2 | 4 | 3
  Cycle 1 Day 1 |  |  | 0.0268 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 0.00358 (83.7) |  | 0.0147 (32.9) | 0.0283 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 0.00258 (45.3) | 0.00380 (102.9) | 0.00628 (108.4)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 2 | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 |  | 0.0415 (21.3) | 0.0167 (37.9) | 0.00261 (66.5) | 0.00820 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 0.0149 (22.0) |  |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 4 | 1
  Cycle 2 Day 1 |  |  | 0.0143 (49.2) |  |  |  | 0.00540 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 0.00226 (52.1) | 0.00306 (55.3) | 0.00700 (NA) — Geometric coefficient of variation was not estimable for a single participant.

21. Secondary Outcome: Part 1: Vss: Volume of Distribution at Steady State for Modakafusp Alfa
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. V(ss) = (dose/AUC)*MRT, where MRT is mean residence time. As per planned analysis, data for this outcome measure was collected and reported dose-wise for each treatment schedule.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/kg
Arm/Group | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.01 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.1 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule A: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.2 mg/kg | Part 1 (Dose Escalation) Schedule B: Modakafusp Alfa 0.3 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 1 (Dose Escalation) Schedule C: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 0.75 mg/kg | Part 1 (Dose Escalation) Schedule D: Modakafusp Alfa 1.5 mg/kg
Number analyzed (Participants) | 0 | 2 | 3 | 3 | 1 | 2 | 1 | 2 | 4 | 3
liters/kg
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 3 | 0 | 2 | 1 | 2 | 4 | 3
  Cycle 1 Day 1 |  |  | 0.104 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 0.0352 (23.4) |  | 0.0575 (26.4) | 0.117 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 0.0329 (32.1) | 0.0390 (27.1) | 0.0536 (24.3)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 2 | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 |  | 0.150 (24.6) | 0.0675 (36.9) | 0.0319 (43.3) | 0.0660 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 0.0624 (14.2) |  |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 4 | 1
  Cycle 2 Day 1 |  |  | 0.0678 (31.1) |  |  |  | 0.0640 (NA) — Geometric coefficient of variation was not estimable for a single participant. | 0.0456 (36.9) | 0.0404 (26.8) | 0.0716 (NA) — Geometric coefficient of variation was not estimable for a single participant.

22. Secondary Outcome: Parts 1, 2 and 3: Percentage of Participants With Positive Anti-drug Antibody (ADA) at Any Scheduled and Unscheduled Post-Baseline Visit
Description: ADA samples scoring equal to or above the cut-point (titer of 75) were defined as ADA positive. Percentages were rounded off to the nearest decimal.
Time Frame: Up to 54.3 months in Part 1; Up to 34.7 months in Part 2; Up to 20.5 months in Part 3
Population: The Immunogenicity-evaluable Analysis Set included participants from the SAS with a baseline assessment and at least 1 postbaseline immunogenicity assessment. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 17 | 6 | 6 | 18 | 7 | 3 | 21 | 7 | 65 | 65
percentage of participants | 41.2 | 83.3 | 83.3 | 66.7 | 57.1 | 66.7 | 61.9 | 14.3 | 52.3 | 61.5

23. Secondary Outcome: Part 1: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved a PR rate or better (sCR + CR + VGPR + PR) during the study as defined by IMWG uniform response criteria. PR: ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. CR: negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow. sCR: CR+normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis, or ≥90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours. Percentages were rounded off to the nearest decimal.
Time Frame: Up to 54.3 months in Part 1
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573 and with measurable disease at baseline. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D
Number analyzed (Participants) | 19 | 8 | 7 | 21
percentage of participants | 15.8 [3.8 to 39.58] | 0 [0.00 to 36.94] | 0 [0.00 to 40.96] | 23.8 [8.22 to 47.17]

24. Secondary Outcome: Parts 1 and 2: Clinical Benefit Rate (CBR)
Description: The CBR was defined as the percentage of participants with a confirmed response of sCR, CR, VGPR, PR, or minimal response (MR) during the study per investigator assessment as defined by IMWG Uniform Response Criteria. PR: ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. CR: negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow. sCR: CR+normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis, or ≥90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours. MR: ≥25% but ≤49% reduction of serum M-protein and reduction in 24-hour urine M-protein by 50% to 89%. Percentages were rounded off to the nearest decimal.
Time Frame: Up to 54.3 months in Part 1; Up to 34.7 months in Part 2
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573 and with measurable disease at baseline. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone
Number analyzed (Participants) | 19 | 8 | 7 | 21 | 8 | 3 | 25 | 25
percentage of participants | 15.8 [3.38 to 39.58] | 0 [0.00 to 36.94] | 0 [0.00 to 40.96] | 38.1 [18.11 to 61.56] | 0 [0.00 to 36.94] | 0 [0.00 to 70.76] | 52.0 [31.31 to 72.20] | 32.0 [14.95 to 53.50]

25. Secondary Outcome: Parts 1 and 2: Disease Control Rate (DCR)
Description: The DCR was defined as the proportion of participants with a confirmed response of sCR, CR, VGPR, PR, MR, or stable disease (SD) during the study per investigator assessment as defined by IMWG Uniform Response Criteria. PR: ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. CR: negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow. sCR: CR+normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis, or ≥90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours. MR: ≥25% but ≤49% reduction of serum M-protein and reduction in 24-hour urine M-protein by 50% to 89%. SD: no known evidence of progressive or new bone lesions if radiographic studies were performed. Percentages were rounded off to the nearest decimal.
Time Frame: Up to 54.3 months in Part 1; Up to 34.7 months in Part 2
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone
Number analyzed (Participants) | 19 | 8 | 7 | 21 | 8 | 3 | 25 | 25
percentage of participants | 57.9 [33.50 to 79.75] | 37.5 [8.52 to 75.51] | 42.9 [9.90 to 81.59] | 61.9 [38.44 to 81.89] | 62.5 [24.49 to 91.48] | 66.7 [9.43 to 99.16] | 64.0 [42.52 to 82.03] | 68.0 [46.50 to 85.05]

26. Secondary Outcome: Parts 1, 2, and 3: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documentation of response PR or better (sCR + CR + VGPR + PR) to the time of disease progression or death, whichever occurs first. PR: ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. CR: negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow. sCR: CR+normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis, or ≥90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours.
Time Frame: Up to 54.3 months in Part 1; Up to 34.7 months in Part 2; Up to 20.5 months in Part 3
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Median (Full Range); unit: months
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 3 | 0 | 0 | 2 | 0 | 0 | 7 | 3 | 6 | 13
months | 2.1 [2.0 to 12.0] |  |  | 7.4 [2.8 to 24.8] |  |  | 24.4 [1.0 to 39.7] | 10.3 [1.0 to 17.6] | NA [2.07 to 13.57] — Median was not reached. | 9.2 [0.76 to 16.82]

27. Secondary Outcome: Parts 1 and 2: Time to Response
Description: Time to response was defined as the time from first dose to the date of first documentation of response (PR or better [sCR + CR + VGPR + PR]) PR: ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. CR: negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow. sCR: CR+normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis, or ≥90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours.
Time Frame: Up to 54.3 months in Part 1; Up to 34.7 months in Part 2
Population: as for outcome 26
Measure: Median (Full Range); unit: months
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone
Number analyzed (Participants) | 3 | 0 | 0 | 5 | 0 | 0 | 12 | 8
months | 1.15 [1.0 to 3.0] |  |  | 1.87 [0.9 to 3.7] |  |  | 1.07 [0.8 to 5.8] | 1.08 [1.0 to 10.0]

28. Secondary Outcome: Parts 1, 2, and 3: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of enrollment until the date of progressive disease (PD) or death due to any cause, whichever occurs first as defined by IMWG Criteria. Per IMWG criteria, PD: serum M-component increase ≥0.5 g/dl or urine M-component increase ≥ 200 mg/24-hour/ difference between involved and uninvolved FLC levels increase >10 mg/dl or bone marrow plasma cell ≥10%/ development of new/ increase in size of existing bone lesions or soft tissue plasmacytoma or development of hypercalcemia.
Time Frame: Up to 54.3 months in Part 1; Up to 34.7 months in Part 2; Up to 20.5 months in Part 3
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573. The FAS included all participants who received at least 1 dose, even an incomplete dose, of modakafusp alfa, in the Part 3 extension cohorts. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 15 | 7 | 6 | 15 | 7 | 2 | 18 | 13 | 43 | 44
months | 2.6 [0.0 to 13.1] | 1.5 [0.2 to 5.4] | 1.4 [0.1 to 6.2] | 3.6 [0.0 to 26.5] | 1.1 [0.5 to 2.3] | 1.4 [0.7 to 1.4] | 8.0 [0.0 to 40.4] | 3.4 [0.0 to 22.7] | 4.1 [0.03 to 15.44] | 5.3 [0.03 to 19.81]

29. Secondary Outcome: Parts 2 and 3: Overall Survival (OS)
Description: The OS was defined as the time from the date of first dose to the date of death due to any cause.
Time Frame: Up to 34.7 months in Part 2; Up to 20.5 months in Part 3
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573. The FAS included all participants who received at least 1 dose, even an incomplete dose, of modakafusp alfa, in the Part 3 extension cohorts. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Median (Full Range); unit: months
Arm/Group | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 18 | 17
months | NA [1.5 to 19.9] — Median was not reached. | NA [1.7 to 15.2] — Median was not reached. | NA [0.5 to 22.3] — Median was not reached. | 3.4 [1.0 to 3.7] | NA [1.08 to 17.25] — Median was not reached. | NA [0.39 to 19.81] — Median was not reached.

30. Secondary Outcome: Part 2: Cmax: Maximum Observed Serum Concentration for Modakafusp Alfa
Time Frame: Schedule C and D: Pre-infusion and at multiple times post-infusion on Day 1 of Cycles 1 and 2: (cycle length was 21 days for Schedule C and 28 days for Schedule D)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg: Participants received modakafusp alfa 0.4 mg/kg infusion, IV, Q3W on Day 1 of each 21-day treatment cycle until treatment discontinuation.
- Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg + Dexamethasone 40 mg: Participants received modakafusp alfa 0.4 mg/kg infusion, IV, and dexamethasone 40 mg, orally, Q3W on Day 1 of each 21-day treatment cycle until treatment discontinuation.
- Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg: Participants received modakafusp alfa 1.5 mg/kg infusion, IV, Q4W on Day 1 of each 28-day treatment cycle until treatment discontinuation.
- Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg + Dexamethasone 40 mg: Participants received modakafusp alfa 1.5 mg/kg infusion, IV, and dexamethasone 40 mg, orally, Q4W on Day 1 of each 28-day treatment cycle until treatment discontinuation.
Arm/Group | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg + Dexamethasone 40 mg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg + Dexamethasone 40 mg
Number analyzed (Participants) | 7 | 3 | 21 | 6
ng/mL
  Cycle 1 Day 1 | 3540 (83.7) | 4330 (23.7) | 32100 (25.4) | 35700 (20.0)
  Cycle 2 Day 1: number analyzed (Participants) | 6 | 3 | 16 | 4
  Cycle 2 Day 1 | 3450 (51.2) | 3870 (26.6) | 34200 (24.6) | 36100 (25.6)

31. Secondary Outcome: Part 2: AUC∞: Area Under the Serum Concentration-time Curve From Time 0 to Infinity for Modakafusp Alfa
Time Frame: as for outcome 30
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg + Dexamethasone 40 mg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg + Dexamethasone 40 mg
Number analyzed (Participants) | 3 | 2 | 19 | 6
h*ng/mL
  Cycle 1 Day 1 | 24900 (77.1) | 42700 (19.2) | 1020000 (89.1) | 1280000 (70.4)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 16 | 3
  Cycle 2 Day 1 | 37200 (35.4) | 43700 (118.5) | 1520000 (60.7) | 2070000 (33.9)

32. Secondary Outcome: Part 2: AUClast: Area Under the Serum Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Modakafusp Alfa
Time Frame: as for outcome 30
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg + Dexamethasone 40 mg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg + Dexamethasone 40 mg
Number analyzed (Participants) | 7 | 3 | 21 | 6
h*ng/mL
  Cycle 1 Day 1 | 40800 (93.6) | 34600 (40.0) | 975000 (90.8) | 1280000 (70.4)
  Cycle 2 Day 1: number analyzed (Participants) | 6 | 3 | 16 | 4
  Cycle 2 Day 1 | 42300 (64.8) | 45600 (74.7) | 1510000 (62.5) | 1650000 (56.3)

33. Secondary Outcome: Part 2: λz: Terminal Disposition Rate Constant for Modakafusp Alfa
Time Frame: as for outcome 30
Population: The PK Analysis Set included participants from the SAS who had sufficient data to calculate at least 1 PK parameter for modakafusp alfa. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis during the specified time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg + Dexamethasone 40 mg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg + Dexamethasone 40 mg
Number analyzed (Participants) | 3 | 2 | 21 | 6
1/h
  Cycle 1 Day 1 | 0.114 (67.0) | 0.111 (31.0) | 0.0478 (63.6) | 0.0468 (62.8)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 16 | 4
  Cycle 2 Day 1 | 0.127 (80.1) | 0.171 (64.0) | 0.0381 (36.9) | 0.0276 (54.4)

34. Secondary Outcome: Part 2: Tmax: Time to Reach the Cmax for Modakafusp Alfa
Time Frame: as for outcome 30
Population: as for outcome 33
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg + Dexamethasone 40 mg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg + Dexamethasone 40 mg
Number analyzed (Participants) | 7 | 3 | 21 | 6
hours
  Cycle 1 Day 1 | 5.70 [4.08 to 7.73] | 3.27 [2.60 to 9.00] | 1.18 [0.93 to 3.00] | 1.68 [1.07 to 6.57]
  Cycle 2 Day 1: number analyzed (Participants) | 6 | 3 | 16 | 4
  Cycle 2 Day 1 | 5.68 [3.88 to 6.68] | 3.30 [1.12 to 9.00] | 1.29 [0.90 to 4.88] | 1.63 [1.10 to 3.00]

35. Secondary Outcome: Part 2: CL: Clearance for Modakafusp Alfa
Description: Clearance is defined as a quantitative measure of the rate at which a drug substance is removed from the body. CL = dose/AUC.
Time Frame: as for outcome 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/kg
Arm/Group | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg + Dexamethasone 40 mg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg + Dexamethasone 40 mg
Number analyzed (Participants) | 3 | 2 | 19 | 6
L/h/kg
  Cycle 1 Day 1 | 0.0160 (77.4) | 0.00937 (19.0) | 0.00147 (89.9) | 0.00119 (67.9)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 16 | 3
  Cycle 2 Day 1 | 0.0107 (35.6) | 0.00912 (118.7) | 0.000995 (61.2) | 0.000737 (36.5)

36. Secondary Outcome: Part 2: Vss: Volume of Distribution at Steady State for Modakafusp Alfa
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. V(ss) = (dose/AUC)*MRT, where MRT is mean residence time.
Time Frame: as for outcome 30
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg + Dexamethasone 40 mg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg + Dexamethasone 40 mg
Number analyzed (Participants) | 3 | 2 | 19 | 6
L/kg
  Cycle 1 Day 1 | 0.114 (32.8) | 0.0646 (4.7) | 0.0260 (67.6) | 0.0276 (16.7)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 16 | 3
  Cycle 2 Day 1 | 0.0779 (32.2) | 0.0501 (41.8) | 0.0289 (39.6) | 0.0260 (13.7)

37. Secondary Outcome: Part 2: T1/2z: Terminal Elimination Phase Half-life for Modakafusp Alfa
Time Frame: as for outcome 30
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa 0.4 mg/kg + Dexamethasone 40 mg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa 1.5 mg/kg + Dexamethasone 40 mg
Number analyzed (Participants) | 3 | 2 | 21 | 6
hours
  Cycle 1 Day 1 | 6.08 (67.0) | 6.22 (31.0) | 14.5 (63.6) | 14.8 (62.8)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 16 | 4
  Cycle 2 Day 1 | 5.46 (80.1) | 4.07 (64.0) | 18.2 (36.9) | 25.1 (54.2)

38. Secondary Outcome: Part 3: Objective Response Rate (ORR) by Investigator Assessment
Description: ORR was defined as the percentage of participants who achieved a PR rate or better (sCR + CR + VGPR + PR) during the study as defined by IMWG uniform response criteria. PR :≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. CR:negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow. sCR: CR+normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry. VGPR:serum and urine M-protein detectable by immunofixation but not on electrophoresis, or ≥90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours. Percentages were rounded off to the nearest decimal.
Time Frame: Up to 20.5 months in Part 3
Population: The FAS included all participants who received at least 1 dose, even an incomplete dose, of modakafusp alfa, in the Part 3 extension cohorts.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 71 | 75
percentage of participants | 32.4 [21.76 to 44.55] | 41.3 [30.08 to 53.30]

39. Secondary Outcome: Part 3: Clinical Benefit Rate (CBR) by IRC and Investigator Assessment
Description: as for outcome 24
Time Frame: Up to 20.5 months in Part 3
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 71 | 75
percentage of participants | 38.0 [26.76 to 50.33] | 48.0 [36.31 to 59.85]

40. Secondary Outcome: Part 3: Duration of Clinical Benefit
Description: Duration of clinical benefit was defined as the time from first documented evidence of confirmed MR or better until the earliest date of a confirmed PD per IMWG, or death among participants who achieve a confirmed MR or better. MR: ≥25% but ≤49% reduction of serum M-protein and reduction in 24-hour urine M-protein by 50% to 89%. Per IMWG criteria, PD: serum M-component increase ≥0.5 g/dl or urine M-component increase ≥ 200 mg/24-hour/ difference between involved and uninvolved FLC levels increase >10 mg/dl or bone marrow plasma cell ≥10%/ development of new/ increase in size of existing bone lesions or soft tissue plasmacytoma or development of hypercalcemia.
Time Frame: Up to 20.5 months in Part 3
Population: The FAS included all participants who received at least 1 dose, even an incomplete dose, of modakafusp alfa, in the Part 3 extension cohorts. Overall number of participants analyzed is the number of participants with events. Participants with no post baseline response assessment were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 27 | 36
months | NA [6.70 to NA] — Due to early termination and low number of participants with post-baseline assessment, median and upper limit of 95% CI was not reached. | 9.2 [4.99 to NA] — Due to early termination and low number of participants with post-baseline assessment, upper limit of 95% CI was not reached.

41. Secondary Outcome: Part 3: Disease Control Rate (DCR) by IRC and Investigator Assessment
Description: as for outcome 25
Time Frame: Up to 20.5 months in Part 3
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 71 | 75
percentage of participants | 74.6 [62.92 to 84.23] | 68.0 [56.22 to 78.31]

42. Secondary Outcome: Part 3: Duration of Disease Control
Description: Duration of disease control was defined as the time from first documented evidence of SD or better until the earliest date of a confirmed PD per IMWG, or death among participants who achieved a SD or better. SD: no known evidence of progressive or new bone lesions if radiographic studies were performed. Per IMWG criteria, PD: serum M-component increase ≥0.5 g/dl or urine M-component increase ≥200 mg/24-hour/ difference between involved and uninvolved FLC levels increase >10 mg/dl or bone marrow plasma cell ≥10%/ development of new/ increase in size of existing bone lesions or soft tissue plasmacytoma or development of hypercalcemia.
Time Frame: Up to 20.5 months in Part 3
Population: The FAS included all participants who received at least 1 dose, even an incomplete dose, of modakafusp alfa, in the Part 3 extension cohorts. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Median (Full Range); unit: months
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 30 | 25
months | 6.5 [0.03 to 14.52] | 5.6 [0.03 to 18.89]

43. Secondary Outcome: Part 3: Time to Progression (TTP) by IRC and Investigator Assessment
Description: TTP was defined as the time from the date of the first dose until the earliest date of confirmed PD per IMWG, or death due to PD. Per IMWG criteria, PD: serum M-component increase ≥0.5 g/dl or urine M-component increase ≥200 mg/24-hour/ difference between involved and uninvolved FLC levels increase >10 mg/dl or bone marrow plasma cell ≥10%/ development of new/ increase in size of existing bone lesions or soft tissue plasmacytoma or development of hypercalcemia.
Time Frame: Up to 20.5 months in Part 3
Population: as for outcome 42
Measure: Median (Full Range); unit: months
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 37 | 39
months | 4.7 [0.03 to 15.44] | 5.5 [0.03 to 19.81]

44. Secondary Outcome: Part 3: Rate of Minimal Residual Disease (MRD) Negativity Status at a Sensitivity of 10^-5 in Participants Achieving CR
Description: MRD negativity rate at a sensitivity of 10^-5 was defined as participants who were MRD negative at a sensitivity of 10^-5 in participants achieving suspected complete response (CR). CR was defined as negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow; in participants for whom only measurable disease is by serum FLC level, normal FLC ratio of 0.26 to 1.65 in addition to CR criteria was required.
Time Frame: Up to 20.5 months in Part 3
Population: The Intent-to-Treat (ITT) Analysis Set included all randomized participants regardless of whether they received study drug or adhered to the assigned dose. Overall number of participants analyzed is the number of participants from ITT analysis set who achieved CR.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

45. Secondary Outcome: Part 3: Duration of MRD Negativity Status at a Sensitivity of 10^-5 in Participants Achieving CR
Description: Duration of MRD negativity (10^-5) was defined as the time from the first MRD negative status (10^-5) to the earliest date of the MRD positive status (10^-5), confirmed PD per IMWG or death.
Time Frame: Up to 20.5 months in Part 3
Population: The ITT Analysis Set included all randomized participants regardless of whether they received study drug or adhered to the assigned dose. Overall number of participants analyzed is the number of participants from ITT analysis set who achieved CR.
Measure: Median (Standard Deviation); unit: months
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 1 | 1
months | NA (NA) — Due to insufficient number of participants the median of duration of MRD negativity could not be accurately obtained. | NA (NA) — Due to insufficient number of participants the median of duration of MRD negativity could not be accurately obtained.

46. Secondary Outcome: Part 3: Percentage of Participants With Treatment -Emergent Adverse Events (TEAEs)
Description: as for outcome 5
Time Frame: Up to 20.5 months in Part 3
Population: as for outcome 38
Measure: Number; unit: percentage of participants
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 71 | 75
percentage of participants | 98.6 | 100

47. Secondary Outcome: Part 3: Percentage of Participants With Serious Treatment-emergent Adverse Events (Serious TEAEs)
Description: AE: any untoward medical occurrence in participants administered pharmaceutical product; untoward medical occurrence does not necessarily have causal relationship with this treatment. AE can therefore be any unfavorable & unintended sign (including abnormal laboratory finding), symptom/disease temporally associated with use of medicinal (investigational) product whether or not it is related to medicinal product. TEAE: any AE either reported for first time or worsening of pre-existing event after first dose of study drug & within 30 days of last administration of study drug. Serious TEAEs: any untoward medical occurrence that: 1) results in death, 2) is life-threatening, 3) requires inpatient hospitalization or prolongation of existing hospitalization, 4) results in persistent or significant disability/incapacity, 5) leads to a congenital anomaly/birth defect in the offspring of the participant or 6) is a medically important event. Percentages were rounded off to the nearest decimal.
Time Frame: Up to 20.5 months in Part 3
Population: as for outcome 38
Measure: Number; unit: percentage of participants
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 71 | 75
percentage of participants | 39.4 | 44.0

48. Secondary Outcome: Part 3: Percentage of Participants With Clinically Significant Laboratory Values
Description: Laboratory values included hematology, chemistry, and urinalysis as interpreted by the investigator.
Time Frame: Up to 20.5 months in Part 3
Population: FAS:all participants who took ≥1 dose,even if incomplete,of TAK-573 in Part 3 extension cohorts.However,clinically significant laboratory values data were not collected&will never be available to present due to issue with report form used for data collection(identified after trial completion).Assessments of clinical significance were not included in report form,making data collection impossible.This issue did not impact participant safety/reliability of study data,particularly primary endpoint.
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 0 | 0

49. Secondary Outcome: Part 3: Number of Participants at Baseline and at Worst Post-baseline Status as Categorized by Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: ECOG performance status was measured at baseline and over time. ECOG performance status was measured on a 6 point scale: Grade 0: Normal activity, Grade 1: Symptoms but ambulatory, Grade 2: In bed <50% of the time, Grade 3: In bed >50% of the time, Grade 4: 100% bedridden, Grade 5: Dead. Reported here is the baseline status and the worst post-baseline status measured. A decrease in grade from baseline indicates an improvement. Only categories for which there was at least 1 participant are reported.
Time Frame: Up to 20.5 months in Part 3
Population: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 68 | 63
Participants
  Baseline: 0; Worst Post-baseline: 0 | 11 | 6
  Baseline: 0; Worst Post-baseline: 1 | 5 | 12
  Baseline: 0; Worst Post-baseline: 2 | 2 | 1
  Baseline: 0; Worst Post-baseline: 3 | 0 | 1
  Baseline: 1; Worst Post-baseline: 0 | 1 | 0
  Baseline: 1; Worst Post-baseline: 1 | 31 | 25
  Baseline: 1; Worst Post-baseline: 2 | 6 | 12
  Baseline: 1; Worst Post-baseline: 3 | 3 | 1
  Baseline: 1; Worst Post-baseline: 4 | 1 | 0
  Baseline: 2; Worst Post-baseline: 2 | 6 | 4
  Baseline: 2; Worst Post-baseline: 3 | 1 | 1
  Baseline: 2; Worst Post-baseline: 4 | 1 | 0

50. Secondary Outcome: Part 3: Health Care Utilization: Length of Hospital Stays
Time Frame: Up to 20.5 months in Part 3
Population: as for outcome 42
Measure: Median (Full Range); unit: days
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 71 | 75
days | 14 [2 to 240] | 11 [1 to 158]

51. Secondary Outcome: Part 3: Percentage of Participants With Neutralizing Antibodies (NAb) at Any Scheduled and Unscheduled Post-Baseline Visit
Description: Percentages were rounded off to the nearest decimal.
Time Frame: Up to 20.5 months in Part 3
Population: Immunogenicity-Evaluable Set Analysis included participants with a baseline assessment and at least 1 post-baseline immunogenicity assessment. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 65 | 65
percentage of participants | 47.7 | 44.6

52. Secondary Outcome: Part 3: Health Care Utilization: Number of Participants With at Least One Medical Encounter
Description: Medical encounters included hospitalizations, emergency room stays, or outpatient visits.
Time Frame: Up to 20.5 months in Part 3
Population: as for outcome 42
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 46 | 57
Participants
  Hospitalizations | 29 | 31
  Emergency Room Stays | 7 | 8
  All Outpatient Visits | 10 | 18

53. Secondary Outcome: Part 3: Patient-reported Outcome (PRO): Change From Baseline to Cycle 9 in Instrument European Organisation for Research and Treatment of Cancer QLQ Questionnaire Multiple Myeloma Module (EORTC QLQ-MY20)
Description: EORTC QLQ-MY20 is a myeloma-specific module developed by the EORTC group specifically to assess quality of life in participants with multiple myeloma. It contains 20 items which can be grouped into a disease symptom subscale (6 items), side effects of treatment subscale (10 items), body image (1 item) and future perspective subscale (3 items). All transformed scale scores range from 0 to 100 with higher scores indicating worse symptoms (Disease Symptoms and Side Effects of Treatment) or better support/functioning (Future Perspective and Body Image).
Time Frame: Baseline, Cycle 9 Day 8 [cycle length was 28 days] (up to 7.7 months)
Population: The PRO Analysis Set included all participants with a baseline and at least one post-baseline measurement of any PRO measure (EORTC QLQ-MY20 or EQ-5D-5L). Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg
Number analyzed (Participants) | 7 | 6
score on a scale
  Disease Symptoms | -7.9 (22.63) | -7.4 (10.93)
  Side Effects of Treatment | 4.7 (11.62) | 7.0 (5.45)
  Body Image | 4.8 (35.63) | 0.0 (21.06)
  Future Perspective | 11.1 (9.06) | 7.4 (34.92)

ADVERSE EVENTS:
Time Frame: Up to 54.3 months in Part 1; Up to 34.7 months in Part 2; Up to 20.5 months in Part 3 and Up to 12.1 months in Japan Lead-in
Description: The SAS included all enrolled participants who received at least 1 dose, even if incomplete, of TAK-573. As pre-planned Adverse Events data was collected and reported "Per Schedule".
Arm/Group | Part 1 (Dose Escalation) Schedule A | Part 1 (Dose Escalation) Schedule B | Part 1 (Dose Escalation) Schedule C | Part 1 (Dose Escalation) Schedule D | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone | Part 3 (Dose Extension): Modakafusp Alfa 120 mg | Part 3 (Dose Extension): Modakafusp Alfa 240 mg | Japan Lead-in: Modakafusp Alfa 60 mg | Japan Lead-in: Modakafusp Alfa 120 mg
All-Cause Mortality (participants affected / at risk) | 15/20 | 6/8 | 6/7 | 8/21 | 3/8 | 1/3 | 5/25 | 6/25 | 19/71 | 20/75 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 8/20 | 6/8 | 2/7 | 13/21 | 1/8 | 1/3 | 7/25 | 9/25 | 28/71 | 33/75 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 20/20 | 8/8 | 7/7 | 21/21 | 8/8 | 3/3 | 24/25 | 24/25 | 70/71 | 74/75 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (Dose Escalation) Schedule A (N=20) | Part 1 (Dose Escalation) Schedule B (N=8) | Part 1 (Dose Escalation) Schedule C (N=7) | Part 1 (Dose Escalation) Schedule D (N=21) | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa (N=8) | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone (N=3) | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa (N=25) | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone (N=25) | Part 3 (Dose Extension): Modakafusp Alfa 120 mg (N=71) | Part 3 (Dose Extension): Modakafusp Alfa 240 mg (N=75) | Japan Lead-in: Modakafusp Alfa 60 mg (N=3) | Japan Lead-in: Modakafusp Alfa 120 mg (N=2)
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 2 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device related bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrophoresis protein abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 2 | 0 | 0
Light chain analysis increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 4 | 0 | 0 | 3 | 4 | 6 | 7 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stupor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (Dose Escalation) Schedule A (N=20) | Part 1 (Dose Escalation) Schedule B (N=8) | Part 1 (Dose Escalation) Schedule C (N=7) | Part 1 (Dose Escalation) Schedule D (N=21) | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa (N=8) | Part 2 (Dose Expansion): Schedule C: Modakafusp Alfa + Dexamethasone (N=3) | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa (N=25) | Part 2 (Dose Expansion): Schedule D: Modakafusp Alfa + Dexamethasone (N=25) | Part 3 (Dose Extension): Modakafusp Alfa 120 mg (N=71) | Part 3 (Dose Extension): Modakafusp Alfa 240 mg (N=75) | Japan Lead-in: Modakafusp Alfa 60 mg (N=3) | Japan Lead-in: Modakafusp Alfa 120 mg (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 5 | 0 | 2 | 3 | 1 | 0 | 3 | 2 | 6 | 11 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 5 | 5 | 3 | 15 | 3 | 3 | 14 | 11 | 31 | 32 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 4 | 1 | 0 | 5 | 3 | 3 | 5 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 1 | 1 | 6 | 1 | 0 | 4 | 4 | 7 | 11 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 8 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 3 | 1 | 0 | 7 | 2 | 7 | 10 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 0 | 3 | 2 | 0 | 1 | 1 | 3 | 2 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 2 | 4 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood uric acid decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 5 | 6 | 0 | 0
Brain fog (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 3 | 4 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 6 | 2 | 0 | 5 | 1 | 7 | 5 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease-mineral and bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 5 | 6 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 2 | 4 | 0 | 0 | 7 | 4 | 12 | 22 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 8 | 14 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 1 | 4 | 3 | 3 | 1 | 6 | 15 | 13 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 7 | 8 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 4 | 1 | 0 | 5 | 5 | 7 | 14 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 5 | 0 | 0 | 0 | 3 | 3 | 4 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 4 | 0 | 0 | 2 | 1 | 4 | 5 | 1 | 0
Fatigue (General disorders) | 8 | 2 | 2 | 8 | 3 | 1 | 7 | 6 | 21 | 29 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 5 | 3 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 5 | 2 | 2 | 7 | 3 | 13 | 11 | 2 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 2 | 5 | 9 | 5 | 2 | 4 | 4 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 7 | 4 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 1 | 0 | 6 | 1 | 0 | 3 | 4 | 2 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 1 | 1 | 5 | 4 | 0 | 9 | 2 | 2 | 6 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2 | 1 | 2 | 1 | 1 | 4 | 5 | 6 | 9 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 4 | 0 | 1 | 2 | 2 | 3 | 6 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 4 | 1 | 3 | 1 | 1 | 4 | 3 | 2 | 4 | 0 | 0
Hypoperfusion (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 0 | 1 | 8 | 2 | 2 | 4 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 3 | 0 | 1 | 2 | 2 | 4 | 3 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 2 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 6 | 3 | 0 | 8 | 3 | 16 | 11 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 2 | 2 | 2 | 1 | 3 | 0 | 4 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 10 | 2 | 5 | 15 | 5 | 3 | 12 | 12 | 18 | 25 | 2 | 1
Lymphocyte count decreased (Investigations) | 9 | 0 | 1 | 11 | 6 | 2 | 7 | 7 | 5 | 6 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 4 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 8 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 7 | 6 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 6 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 0 | 7 | 2 | 0 | 7 | 5 | 11 | 22 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 4 | 5 | 16 | 5 | 3 | 18 | 15 | 48 | 55 | 3 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 5 | 1 | 0 | 0
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 2 | 0 | 2 | 2 | 5 | 5 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 6 | 13 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 4 | 4 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 4 | 1 | 1 | 2 | 2 | 2 | 6 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 7 | 3 | 8 | 16 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 3 | 4 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 4 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 8 | 6 | 16 | 6 | 3 | 19 | 20 | 52 | 63 | 2 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 3 | 0 | 1 | 2 | 5 | 6 | 12 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 7 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 3 | 0 | 1 | 3 | 4 | 3 | 6 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 6 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to discontinuation of development of modakafusp alfa for strategic reasons. The November 7 2024 data cut comprises the final full dataset for safety and efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT03215030/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03215030/SAP_001.pdf